CLINICAL TRIAL: NCT00425971
Title: A Phase 1, Double-Blind, Randomized, Placebo-Controlled, Dose-Escalating Safety Study of BMEC-1217B, in Healthy Volunteers
Brief Title: Safety Study of Anti-Asthma Agent BMEC-1217B
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medigreen Biotechnology Corp. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ITRI-BEL1217B-CP002
Record Dates: First submitted 2007-01-23; First posted 2007-01-24 (Estimated); Last update posted 2008-09-04 (Estimated); Status verified 2008-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

INTERVENTIONS:
Drug: BMEC-1217B

SUMMARY:
BMEC-1217B is an abbreviated version of an old Chinese formulation. The ratio of each component was adopted by the sponsor following the observation that BMEC-1217B prepared from this ratio resulted in best pharmacological profile and in vitro bioactivities.

BMEC-1217B was studied for the pharmacological activity on the release of cysteinyl leukotrienes, IL-4 and TNF-alpha in vitro and the airway hyperreactivity. The result indicated that BMEC-1217B can inhibit the synthesis of several key pro-inflammatory mediators involved in the pathophysiology of allergic asthma and can also improve lung function in a mouse model of allergic asthma.

The purpose of this study is to evaluate the safety and tolerability of increasing dose of BMEC-1217B when administered orally in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Nonsmoking healthy adults between 20 and 40 years old.
2. Determined to be in good health based on medical history, clinical laboratory test values within normal range. Body weight within 20% of the ideal body weight [(height - 80) x 0.7].
3. No recent history of drug or alcohol abuse within one year prior to study enrollment
4. Signed informed consent form.

Exclusion Criteria:

1. Has any condition that interferes with the ability of the subject to comply with the requirements of the study.
2. Has known allergy to the study drug.
3. Has an acute illness or surgery within 28 days prior to study enrollment
4. Has participated in other investigational trials within 28 days prior to study enrollment.
5. Has taken prescription medication and/or over-the-counter medication*4 and/or botanical medications within 28 days prior to study enrollment.
6. Has alcohol and caffeine consumption within 24 hours prior to the administration of study drug.
7. Has evidence of significant renal, cardiovascular, hepatic, hematopoetic, neurological, pulmonary or gastrointestinal pathology, or any other medical reason or disease that might interfere with the study objectives, as determined by the investigator.
8. Has donation or receive of more than 450 mL of blood within 28 days prior to the study enrollment.
9. Female subjects of child bearing potential who are pregnant, nursing, do not agree to practice effective birth control during the time period from 14 days before administration of study drug to 28 days after administration of study drug, or with irregular or abnormal menstruation.
10. Clinically significant deviation from normal physical examination findings that, in the principal investigator's judgment, may interfere with the study evaluation or affect subject safety.
11. Test positive for HIV, HBV or HCV
12. Test results indicate liver function failure
13. Has been diagnosed with Diabetes Mellitus

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2008-07

CONTACTS AND LOCATIONS:
Overall Officials: Horng-Chin Yan, M.D., Ph.D., Principal Investigator — Tri-Service General Hospital, Taipei, Taiwan
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan